CLINICAL TRIAL: NCT01215552
Title: A PET Study: Single-dose, Open-label Study of the Inhibition of [11C]R-rolipram Binding to Brain Phosphodiesterase - 4 (PDE-4) by HT-0712
Brief Title: Study of the Inhibition of [11C]R-rolipram Binding to Brain Phosphodiesterase - 4 (PDE-4) by HT-0712
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The experimental design was not sufficient to answer the proposed questions. A new study design is now being considered.
Sponsor: Dart NeuroScience, LLC (Industry)
Responsible Party: Dr. Philip Perera, MD, Helicon Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HT-0712-006; BNL IRB #444 (Other: Brookhaven National Laboratory)
Record Dates: First submitted 2010-09-24; First posted 2010-10-06 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Elderly Volunteers
MeSH Terms: interventions — HT-0712

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HT-0712 (Experimental)
  Interventions: Drug: HT-0712

INTERVENTIONS:
Drug: HT-0712 — A range of single oral dose levels will be explored, utilizing 5mg and 25mg strength capsules

SUMMARY:
This Positron Emission Tomography (PET) imaging study is designed to explore the relationship between HT-0712 dose level and inhibition of brain phosphodiesterase-4 activity, in order to optimize the dosage regimens utilized in subsequent trials.

DETAILED DESCRIPTION:
The objective of this project is to demonstrate the inhibition of human brain PDE4 by HT-0712, by measuring the inhibition of [11C]R-rolipram binding, a radiotracer which also binds to and inhibits PDE4. Plasma samples will be drawn to determine if there is a relationship between plasma pharmacokinetics of HT-0712 and its pharmacodynamic effect, as determined through the inhibition of [11C]R-rolipram binding in the brain.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy, elderly, non-smoking men and post-menopausal women
* Ability to give informed consent

Main Exclusion Criteria:

* Current or history of uncontrolled hypertension, major depression, Parkinson's disease, stroke and diabetes.
* Physical or behavioral conditions that may alter brain function

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
PET measurement of HT-0712 inhibition of [11C]R-rolipram binding | 1 day
  To demonstrate Central Nervous System (CNS) exposure and dose-related inhibition of [11C]R-rolipram binding in brain regions of interest by HT-0712 when compared to baseline [11C]R-rolipram binding in the same individual.

SECONDARY OUTCOMES:
Brain uptake of [11C]R-rolipram, as determined by PET imaging, associated with both maximal plasma concentration of HT-0712 (Tmax) and overall plasma level exposure (AUC) following administration of different dose levels of HT-0712. | 1 day
  Time-activity curves and plasma AUC will be assessed for [11C]R-rolipram at baseline and at 4-hours post oral administration of HT-0712.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Perera, MD, Study Director — Dart NeuroScience, LLC
Locations (1):
- Brookhaven National Laboratory, Upton, New York, United States